CLINICAL TRIAL: NCT04718987
Title: Potency pReservation In Prostate cAncer Patients Treated With UltraSound-guided Low-dose Rate Brachytherapy
Acronym: PRIAPUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRIAPUS
Record Dates: First submitted 2020-11-16; First posted 2021-01-22 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: Brachytherapy; Radiation; Low Dose Rate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm clinical trial to enroll a total of 10 low- or favourable intermediate-risk prostate cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate Cancer Patients (Experimental): Low- or favourable intermediate-risk prostate cancer patients
  Interventions: Radiation: Low dose rate (LDR) brachytherapy

INTERVENTIONS:
Radiation: Low dose rate (LDR) brachytherapy — Low dose rate (LDR) brachytherapy is a type of radiation treatment where doctor places the radioactive implants (seeds) inside patient's prostate gland and these seeds emits low dose radiation over a certain period of time. During low-dose-rate brachytherapy, a continuous low dose of radiation is released over time -from several hours to several days.

SUMMARY:
The purpose of this study is to develop and evaluate a Magnetic Resonance (MR) fusion 3D Ultrasound (US) guided Low dose rate (LDR) brachytherapy technique that significantly spares prostatic neurovascular bundles (a bundle of nerves and vessels that run beside the prostate) and penile bulb (base of the penis), while still trying to effectively treat the prostate cancer.

DETAILED DESCRIPTION:
Low dose rate (LDR) brachytherapy is an excellent treatment strategy for patients with prostate confined cancers, achieving high curative rates. However, LDR brachytherapy has been linked with long-term erectile dysfunction (ED), with a broad range of reported incidence in the literature.

The pathophysiology associated with ED is complex and variable among different prostate cancer treatment strategies. In the post radical prostatectomy (RP) setting, ED is usually an immediate phenomenon and associated with neuropraxia caused by trauma and inflammation (Nandipati 2006). On the contrary, external beam radiotherapy (EBRT) related ED frequently occurs between 6-24 months and is believed to be vasculogenic in nature and caused by veno-vascular luminal occlusion (Mulhall et al. 2005) that culminates into fibrosis of the corporal tissue. In the post brachytherapy setting, seems plausible that a combination of both nerve and vascular damage are involved in the ED pathogenesis as erectile scores seem to reduce in the first months post implant (likely due to trauma) followed by a subsequent recovery and then, a gradual decline (Mabjeesh 2005).

Despite a more complex pathophysiology, rates of ED post LDR brachytherapy seem to be lower than post EBRT or RP treatment (Crook 2010, Putora 2015). This may be associated with a significantly lower degree of trauma to the surrounding healthy tissue compared with trauma caused by RP and a more conformal dose around the prostate when contrasted with EBRT. In this regard, brachytherapy delivers a lesser dose to important structures previously correlated with an erectile function such as the internal pudendal artery (IPA), penile bulb, corpus cavernosum and possibly the neurovascular bundle.

Currently, some strategies have been developed in an attempt to minimize ED post radiotherapy. In the POTEN-C clinical trial (NCT03525262), 120 patients are being randomized to stereotactic ablative radiotherapy with or without neurovascular sparing (neurovascular bundle, IPA and penile bulb/corpus carvenosum) with ED as the primary endpoint. Although the concept is intriguing, LDR brachytherapy has superior dose conformality and hence, a better chance to reduce radiation dose to the surrounding structures involved in the erectile function while still effectively treating the prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed adenocarcinoma of the prostate
* NCCN-defined low- or favourable intermediate-risk prostate cancer patients
* All pathological cores confined to one lobe of the prostate (minimum of 12 cores sampled), unless a recent multiparametric prostate MR-scan (mpMR) (with < 6 months from the enrollment date) indicates a dominant intra-prostatic lesion (DIL) located at the prostatic lobe where a higher number of cores and Gleason score was found positive. PIRADS v2 score 3-5 lesions are considered DILs.
* No or mild erectile function impairment (score ≥18 in International Index of Erectile Function- 5 [IIEF-5] without PDE-5 inhibitor assistance)
* Sexually active
* No contraindications to prostate LDR brachytherapy

Exclusion Criteria:

* Core positivity in both lobes of the prostate with no DIL detected on mpMR
* mpMR suggesting presence of DILs in both lobes of the prostate
* Contraindications to receiving a MR-scan
* Medically unfit for general and/or spinal anesthesia
* IPSS score > 15
* Inflammatory bowel disease
* Prior abdominal-perineal resection
* Presence of distant metastases and/or nodal disease
* Older than 75 years of age
* Use of cytoreductive prostate treatment (including 5 alpha-reductase inhibitors)
* NCCN-defined unfavourable intermediate or high-risk prostate cancer
* Signs of extra-capsular extension or seminal vesicle involvement on MR-scan
* Prior TURP
* > 3mm of median lobe protrusion to bladder measured in mpMR (Roeloffzen 2011)
* Prior RT to the pelvis
* Significant artifact on MR-Scan (e.g. caused by hip prosthesis)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male only because this study trying to preserve the Penis erection in patients undergoing Radiation treatment for their prostate cancer.
Enrollment: 10 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients receiving this experimental brachytherapy technique and achieving acceptable dose distribution at 1-month post-implant. | 1 month after intervention
  Acceptable dose distribution is defined as:
  1. Target volume (Prostate, excluding a 5 mm expansion of the Neurovascular bundle) D90 ≥ 140 Gy
  2. Contralateral neurovascular bundle median dose ≤ 50 Gy
  3. Prostatic bulb D10 dose ≤ 50 Gy (Chasseray 2019)
  4. Urethra D30 < 130% of the prescription dose

SECONDARY OUTCOMES:
Number of patient with preserved erectile function Erectile Function (IIEF) >= 18) | 1, 6, 12, 18, 24, 36, 48, 60 months post intervention
  The IIEF classifies the severity of ED into five categories stratified by score
  * No ED.26-30
  * Mild.22-25
  * Mild to moderate.17-21
  * Moderate.11-16
  * Severe.6-10
Post-procedure PSA dynamic | 6, 12, 18, 24, 36, 48, 60 months post intervention
  PSA curve post procedure
Acute and long-term GU and GI toxicity | 1, 6, 12, 18, 24, 36, 48, 60 months post intervention
  Evaluate acute and long-term G3 or larger toxicity based on NCI-CTCAE 5.0 score system. Grade 1 to Grade 5. Higher the grade more severe is the toxicity.
Biochemical failure | 1, 6, 12, 18, 24, 36, 48, 60 months post intervention
  Biochemical failure will be assessed according to the Phoenix criteria (nadir + 2.0ng/mL)
Local recurrence | Until study completion with 5 years of follow up
  To assess the rate of biopsy-proven local recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Mendez, MD, Principal Investigator — London Health Sciences Centre- London Regional Cancer Program
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulhall J, Ahmed A, Parker M, Mohideen N. The hemodynamics of erectile dysfunction following external beam radiation for prostate cancer. J Sex Med. 2005 May;2(3):432-7. doi: 10.1111/j.1743-6109.2005.20362.x. PMID 16422876
- [Background] Mabjeesh N, Chen J, Beri A, Stenger A, Matzkin H. Sexual function after permanent 125I-brachytherapy for prostate cancer. Int J Impot Res. 2005 Jan-Feb;17(1):96-101. doi: 10.1038/sj.ijir.3901271. PMID 15510186
- [Background] Putora PM, Engeler D, Haile SR, Graf N, Buchauer K, Schmid HP, Plasswilm L. Erectile function following brachytherapy, external beam radiotherapy, or radical prostatectomy in prostate cancer patients. Strahlenther Onkol. 2016 Mar;192(3):182-9. doi: 10.1007/s00066-015-0928-x. Epub 2015 Dec 28. PMID 26713323
- [Background] Chasseray M, Dissaux G, Bourbonne V, Boussion N, Goasduff G, Malloreau J, Malhaire JP, Fournier G, Tissot V, Pradier O, Valeri A, Schick U. Dose to the penile bulb and individual patient anatomy are predictive of erectile dysfunction in men treated with 125I low dose rate brachytherapy for localized prostate cancer. Acta Oncol. 2019 Jul;58(7):1029-1035. doi: 10.1080/0284186X.2019.1574981. Epub 2019 Feb 14. PMID 30761939
- [Background] Sun Y, Qiu W, Yuan J, Romagnoli C, Fenster A. Three-dimensional nonrigid landmark-based magnetic resonance to transrectal ultrasound registration for image-guided prostate biopsy. J Med Imaging (Bellingham). 2015 Apr;2(2):025002. doi: 10.1117/1.JMI.2.2.025002. Epub 2015 Jun 24. PMID 26158111
- [Background] Crook JM, Gomez-Iturriaga A, Wallace K, Ma C, Fung S, Alibhai S, Jewett M, Fleshner N. Comparison of health-related quality of life 5 years after SPIRIT: Surgical Prostatectomy Versus Interstitial Radiation Intervention Trial. J Clin Oncol. 2011 Feb 1;29(4):362-8. doi: 10.1200/JCO.2010.31.7305. Epub 2010 Dec 13. PMID 21149658